CLINICAL TRIAL: NCT04799535
Title: Quantitative Microvasculature Imaging for Breast Cancer Detection and Monitoring
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-003028; NCI-2021-01733 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-003028 (Other: Mayo Clinic Institutional Review Board); R01CA239548 (NIH)
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma; Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Observational (ultrasound): AIM 1: Participants undergo a breast ultrasound over 15 minutes.
  AIM 2: Participants undergo breast ultrasounds over 15 minutes before starting the chemotherapy and/or endocrine therapy, 2 months after start of chemotherapy and/or endocrine therapy, and after the completion of chemotherapy and/or endocrine therapy before surgery. Participants may also undergo breast ultrasounds at 2 weeks after start of chemotherapy and/or endocrine therapy and 1 month after start of chemotherapy and/or endocrine therapy.
  AIM 3: Patients with suspicious breast masses or known breast cancer who are scheduled for axillary lymph node biopsy undergo ultrasound over 15 minutes at the same visit of the breast mass study.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Undergo breast ultrasound

SUMMARY:
This study evaluates the effectiveness of a breast ultrasound method for the diagnosis of breast cancer. Diagnostic procedures, such as breast ultrasound, may help find and diagnose breast cancer, and may help measure a patient's response to earlier treatment. The purpose of this research is to test the effectiveness of a new investigational breast ultrasound method to detect an abnormality in the breast, and assess response to breast cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the diagnostic performance of the proposed method in a population of pre-biopsy patients with suspicious breast masses and correlate the proposed method results with pathology as the gold standard.

II. Assess and predict the response to preoperative chemotherapy and/or endocrine therapy in breast cancer patients using the proposed method and compare the results to magnetic resonance imaging (MRI) as control and surgical pathology for pathological complete response (PcR).

III. Determine the diagnostic performance of the proposed method in identifying metastatic axillary lymph node in patients with suspected or known breast cancer lesions; correlate the results with pathology as the gold standard.

OUTLINE:

AIM 1: Participants undergo a breast ultrasound over 15 minutes.

AIM 2: Participants undergo breast ultrasounds over 15 minutes before starting the chemotherapy and/or endocrine therapy, 2 months after start of chemotherapy and/or endocrine therapy, and after the completion of chemotherapy and/or endocrine therapy before surgery. Participants may also undergo breast ultrasounds at 2 weeks after start of chemotherapy and/or endocrine therapy and 1 month after start of chemotherapy and/or endocrine therapy .

AIM 3: Patients with suspicious breast masses or known breast cancer who are scheduled for axillary lymph node biopsy undergo ultrasound over 15 minutes at the same visit of the breast mass study.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: Patient volunteers, ages >= 18 with suspicious breast masses scheduled for breast biopsy, or at least two weeks or more after breast biopsy
* AIM 2: Patient volunteers, ages >= 18 who have biopsy proven breast cancer and are going under neoadjuvant chemotherapy and/or endocrine therapy had their baseline MRI and/or ultrasound

Exclusion Criteria:

* Patients with breast implants or any condition that does not allow proper use of ultrasound (US)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers for Aim 1 are without a history of mastectomy or implants, and at least a single suspicious breast mass that is scheduled for biopsy. Volunteers for Aim 2 have biopsy proven breast cancer and are scheduled for chemotherapy and/or endocrine therapy.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2027-11-29 (Estimated); Study Completion 2027-11-29 (Estimated)

PRIMARY OUTCOMES:
Specificity of ultrasound in detection of breast cancer | Up to study completion, an average of 1 year
  Will be reported including 95% confidence intervals derived from the cross-validation procedure.

SECONDARY OUTCOMES:
Accuracy in prediction of treatment response | Up to study completion, an average of 1 year
  Morphological parameters of the lesion's microvasculature will be assessed at each visit. Correlation between changes in the morphological parameters and the clinical measure of lesion size will be assessed. Analyses will be done by time periods separately, change from pre-chemotherapy to halfway through chemotherapy and again from pre to post-chemotherapy. The diagnostic accuracy estimates will be reported along with 95% confidence interval. Univariate associations between changes in microvasculature parameters assessments during a time period with the magnetic resonance imaging (MRI) assessment for change in the same time period will be assessed using logistic regression, reporting the odds ratio and 95% confidence interval. Multi-variable logistic regression will be used to assess independent associations of change in assessments with MRI assessment for change. T-tests will be used to compare microvasculature information between chemotherapy responders and non-responders.

OTHER OUTCOMES:
Specificity of ultrasound in prediction of NUMMA parameters - tortuosity | Up to study completion, an average of 1 year
  The diagnostic accuracy of the NUMMA parameters, such as tortuosity will be assessed using an automated quantification tool. Logistic regression models will examine these collective parameters as predictors of metastatic axillary lymph node in breast cancer patients. Area under the receiver operating characteristic curve (area under the curve) will be examined for univariate and multivariable models. Statistical evaluation of the performance of 2 dimensional (D) and 3D images will be performed with the McNemar's test separately for metastatic and reactive lymph nodes.
Specificity of ultrasound in prediction of NUMMA parameters - vessel diameter | Up to study completion, an average of 1 year
  The diagnostic accuracy of the NUMMA parameters, such as vessel diameter will be assessed using an automated quantification tool. Logistic regression models will examine these collective parameters as predictors of metastatic axillary lymph node in breast cancer patients. Area under the receiver operating characteristic curve (area under the curve) will be examined for univariate and multivariable models. Statistical evaluation of the performance of 2 dimensional (D) and 3D images will be performed with the McNemar's test separately for metastatic and reactive lymph nodes.
Specificity of ultrasound in prediction of NUMMA parameters - numbers of vessel segments | Up to study completion, an average of 1 year
  The diagnostic accuracy of the NUMMA parameters, such as numbers of vessel segments will be assessed using an automated quantification tool. Logistic regression models will examine these collective parameters as predictors of metastatic axillary lymph node in breast cancer patients. Area under the receiver operating characteristic curve (area under the curve) will be examined for univariate and multivariable models. Statistical evaluation of the performance of 2 dimensional (D) and 3D images will be performed with the McNemar's test separately for metastatic and reactive lymph nodes.
Specificity of ultrasound in prediction of NUMMA parameters - vessel density | Up to study completion, an average of 1 year
  The diagnostic accuracy of the NUMMA parameters, such as vessel density will be assessed using an automated quantification tool. Logistic regression models will examine these collective parameters as predictors of metastatic axillary lymph node in breast cancer patients. Area under the receiver operating characteristic curve (area under the curve) will be examined for univariate and multivariable models. Statistical evaluation of the performance of 2 dimensional (D) and 3D images will be performed with the McNemar's test separately for metastatic and reactive lymph nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Alizad, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials